CLINICAL TRIAL: NCT03456817
Title: A Phase 2, Open-label Study to Evaluate Graft-vs-host Disease Prophylaxis With High Dose Thymoglobulin, Methotrexate, and Low-dose Cyclosporine in Comparison to Historical/Concurrent Controls Who Received Low Dose Thymoglobulin, Methotrexate, and High-dose Cyclosporine
Brief Title: HIgh Dose Thymoglobulin Instead of Cyclosporine With a Low Dose of Thymoglobulin for GVHD Prophylaxis
Acronym: ATG2017
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow patient accrual and appearance of a toxicity
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG2017
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Graft-versus-host-disease; Relapse
MeSH Terms: conditions — Graft vs Host Disease; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm - High dose ATG, Low dose CSA (Experimental): High dose ATG will be infused on days -4, -3, -2, -1 and 0. Before each infusion of ATG (thymoglobulin), patient will receive medications preventing side effects from the ATG, including diphenhydramine (Benadryl), an antipyretic (ibuprofen or acetaminophen) and methylprednisolone (Solumedrol). The high dose ATG will be given into patient's vein via central venous catheter. Each infusion of ATG will take 4-8 hours. CSA (cyclosporine A) will be given from day 21. Standard dose methotrexate will be given.
  Interventions: Drug: Treatment Arm - high dose ATG
- Control Arm - Standard of care (Other): Low dose ATG (thymoglobulin) will be infused on days -2, -1 and 0, and CSA (cyclosporine A) will be given from day -1 through day 84. Standard dose methotrexate will also be given.
  Interventions: Drug: Control Arm - standard of care

INTERVENTIONS:
Drug: Treatment Arm - high dose ATG — Patients agreeing to high dose ATG will be treated with 2 mg/kg daily on days -4 to 0. On days -4, -3 & -2, ATG will be infused after fludarabine & busulfan infusion. ATG will be infused over a minimum of 6 hrs on day -4 & over at least 4 hrs on days -3, -2, -1 & 0. Dose is based on actual body wt, & rounded to nearest vial-Thymoglobulin is supplied in 25 mg vials, except if rounding would result in >5% difference from calculated dose. Foothills Medical Center Unit 57 standard practice followed for ATG infusion. ATG premeds include methylprednisolone, diphenhydramine, and an antipyretic. Meperidine 25-50 mg IVPB every 4 hours will be given as needed for rigors. MTX is given 15 mg/m2 IV on day +1 & 10 mg/m2 on days +3, +6 & +11 posttransplant. First dose of methotrexate is given on day +1, at least 24 hrs following end of infusion of stem cell product.
  Arms: Treatment Arm - High dose ATG, Low dose CSA
Drug: Control Arm - standard of care — The historical controls will have received and the concurrent controls will receive our standard GVHD prophylaxis, ie, ATG 4.5 mg/kg i.v. (0.5 mg/kg on day -2, 2.0 mg/kg on day -1 and 2.0 mg/kg on day 0), MTX (15 mg/m2 i.v. on day 1 and 10 mg/m2 i.v. on days 3, 6 and 11) and CSA (2.5 mg/kg twice a day i.v. starting from day -1, adjusting dose to target trough plasma CSA levels of 200-400 microg/L, switching to oral formulation before discharge from peritransplant hospitalization, targeting the trough plasma levels of 200-400 microg/L until day 56, and tapering to zero between day 56 and 84).
  Arms: Control Arm - Standard of care

SUMMARY:
The purpose of this study is to find out whether compared to our standard low dose ATG with CSA, the high dose ATG with low-dose CSA minimizes the chances of relapse and chronic GVHD, without increasing the chances of other transplant complications.

DETAILED DESCRIPTION:
There are a number of complications of allogeneic hematopoietic cell transplantation.

The main complications are:

* Relapse (leukemia or leukemia-like disease returning). This usually leads to death.
* Acute graft-versus-host disease (GVHD). This may lead to death.
* Chronic GVHD. This may lead to poor quality of life long-term.

This study is being done to minimize the chances of patients getting relapse and chronic GVHD, without increasing the chances of getting acute GVHD.

At this time, the standard of care approach to treat this condition would be with:

* Low dose thymoglobulin (ATG), given on Day -2, -1 and 0.
* Cyclosporin (CSA), given from Day -1 through to Day 84.
* Methotrexate, given on Days 1, 3, 6 and 11

CSA reduces the chances of getting acute GVHD, but it does not reduce the chances of getting chronic GVHD and increases the chances of getting relapse. ATG reduces both acute and chronic GVHD, and does not increase relapse.

In this study, high dose ATG will be given on days -4, -3, -2, -1 and 0 (instead of only on days -2, -1 and 0), CSA will be given only from day 21 through 84 (instead of from day -1 through 84), and the routine dose of methotrexate (unchanged) will be given. We think that this may lead to better outcomes.

Patients will be followed per standard practice of the Alberta Blood and Marrow Transplant Program for the development of acute and chronic GVHD, and for relapse.

Patients will also be asked to complete a quality of life questionnaire 2 years after the transplant to assess how their treatment and illness affects their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. First allogeneic HCT, performed for a hematologic malignancy, using filgrastim-mobilized peripheral blood stem cells (PBSC).
2. Conditioning with fludarabine 50 mg/m2 daily on day -6 to -2, busulfan approximately 3.2 mg/kg daily on day -5 to -2 with PK adjustment (target AUC of 3750 uM*min/L) and total body irradiation (TBI) 2 Gy x 2 given typically on day -1 and/or day 0 (before graft infusion), ie, our standard myeloablative conditioning.79 Dose and schedule adjustments per Investigator discretion are permitted.
3. Planned GVHD prophylaxis with our standard of low-dose ATG (4.5 mg/kg) + MTX + high-dose CSA.
4. HLA matched sibling donor, or ≥7/8 HLA allele-matched unrelated donor (maximum 1 allele mismatch at HLA-A, B, C, or DRB1).
5. Age >17 years.

Exclusion Criteria:

1. Nonmyeloablative conditioning.
2. Cord blood or marrow graft.
3. Myelofibrosis being the primary indication for HCT.
4. Previous autologous or allogeneic HCT.
5. Total Bilirubin >1.5-fold above upper normal limit (UNL), ALT >2.0-fold above UNL, or alkaline phosphatase >2.5-fold above UNL.
6. HIV positive by a serologic test that includes detection of both antibody and antigen)
7. Increased risk of tuberculosis, defined as patient requiring an anti-tuberculosis drug peritransplant. All patients with a history of tuberculosis (active or latent) or contact with a person with active tuberculosis will be evaluated by an infectious disease specialist to determine whether treatment or prophylaxis of tuberculosis with an anti-tuberculosis drug peritransplant is needed. The infectious disease specialist will order tests (eg, Mantoux tuberculin skin test or interferon gamma release test) as needed to arrive at the decision on whether an anti-tuberculosis drug peritransplant is needed.
8. High risk of cytomegalovirus (CMV) disease or recurrent CMViremia based on donor negative AND recipient positive CMV serostatus.2 If recipient serostatus was determined since the presentation of his/her hematologic malignancy more than once and the results are discrepant, the determination performed >4 weeks after a transfusion of platelets or plasma (or before transfusions of platelets or plasma were initiated) is considered valid. If unclear, the CMV serostatus determination will be at the discretion of the treating Investigator
9. High risk of PTLD based on donor positive AND recipient negative Epstein-Barr virus (EBV) serostatus (EBNA1 or VCA IgG)80
10. Hypersensitivity to rabbit blood protein, Thymoglobulin or a Thymoglobulin excipient.
11. Severe obesity, defined as body mass index ≥40 kg/m2.81 The reason is that obese patients are at risk of achieving a high ATG area under the time vs concentration curve (AUC).82 This could lead to substantial toxicity (e.g., death due to an infection) when using the studied high dose (10 mg/kg) of ATG.
12. Contraindication to methotrexate:

    1. Hypersensitivity to methotrexate or to any ingredient in the formulation or component of the container.
    2. Females of childbearing potential who are pregnant, breastfeeding or unwilling to use adequate contraception from the time of enrolment until at least day 100 posttransplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
moderate/severe chronic GVHD- and relapse-free survival (cGFRS) at 2 years post transplant | 2 years
  cGRFS will be compared between the study patients and the historical/concurrent controls using a Cox proportional hazards model to determine if administering high dose ATG + MTX and low dose CSA will be associated with improved cGRFS compared to historical/concurrent controls (4.5 mg/kg ATG + MTX + CSA).

SECONDARY OUTCOMES:
quality of life | approximately 2 years (21 to 27 months) post transplant
  each scale (domain) of the short form-36 (SF36) questionnaire will be compared between the high dose ATG group and the control group using Mann-Whitney-Wilcoxon signed rank test to determine if quality of life (QOL) at 2 years posttransplant will be better in the high dose ATG patients compared to the controls (due to the reduction of cGVHD).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Storek, MD, Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Centre/Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada